CLINICAL TRIAL: NCT01770990
Title: Randomized Trial of Telephone-Based Psychotherapy for Depression With and Without Adjunctive Supportive Mail
Brief Title: Trial of Telephone-based Psychotherapy for Depression With and Without Adjunctive Supportive Mail
Acronym: Tel-PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01KQ1002B-TP7-Tel-PT
Record Dates: First submitted 2013-01-08; First posted 2013-01-18 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Depression
Keywords: depression; telephone-based psychotherapy; cognitive-behavioral psychotherapy; manualized psychotherapy; telephone counseling; telephone psychological treatment; telephone-administered therapy; low-intensity treatment; motivational mail; reminder; letter
MeSH Terms: conditions — Depression | interventions — NFKBIZ protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tel-PT without mail (Active Comparator): Telephone-based psychotherapy (1 personal session, 8-10 telephone sessions, educational materials and monitoring questionnaires) without additional motivating letters.
  Interventions: Behavioral: Tel-PT without mail
- Tel-PT including mail (Experimental): Telephone-based psychotherapy (1 personal session, 8-10 telephone sessions, educational materials and monitoring questionnaires) with an additional motivating letter after every telephone session.
  Interventions: Behavioral: Tel-PT including mail

INTERVENTIONS:
Behavioral: Tel-PT including mail — Patients receive telephone-based psychotherapy and one letter after each telephone session.
  Arms: Tel-PT including mail
Behavioral: Tel-PT without mail — Patients receive telephone-based psychotherapy without additional letters.
  Arms: Tel-PT without mail

SUMMARY:
This study aims to compare the effectiveness of two telephone-based psychotherapy (Tel-PT) interventions for patients with mild to moderate depression. Both interventions consist of one personal session and weekly to bi-weekly 8-10 telephone sessions with a licensed cognitive-behavioral psychotherapist accompanied by the study of educational materials and the completion of regular monitoring questionnaires (total treatment duration: approximately 3 months). Patients are randomized into one of two conditions: Patients in the condition "Tel-PT including mail" additionally receive a motivating letter from their psychotherapist after each telephone session, while patients in the condition "Tel-PT without mail" receive no further interventions. Patients refusing to be randomized are to be assigned to the condition "Tel-PT without mail". This study takes place within a larger study evaluating a stepped care model for depression (01KQ1002B-TP7).

DETAILED DESCRIPTION:
The study aims to compare the effectiveness of two telephone-based psychotherapy (Tel-PT) interventions for patients with mild to moderate depression. Patients are randomized into one of two conditions: Patients in the condition "Tel-PT including mail" additionally receive a motivating letter from their psychotherapist after each telephone session, while patients in the condition "Tel-PT without mail" receive no further interventions. Patients refusing to be randomized are to be assigned to the condition "Tel-PT without mail". This study takes place within a larger study evaluating a stepped care model for depression (01KQ1002B-TP7).

In both conditions, patients are referred to telephone-based psychotherapy by their general physician within the framework of the larger study. Both intervention programs are based on the translated and adapted German version of a depression-specific program developed by researchers in Seattle. Both include psycho-educational materials (patient workbook and therapist manual) and comprise 1 personal session, 8 to 10 telephone contacts (20 to 40 minutes) carried out weekly and in some cases bi-weekly, as well as up to 2 maintenance therapy telephone sessions for patients responding well to telephone-based psychotherapy (see monitoring process below). Both programs have a duration of approximately 3 months and follow a cognitive-behavioral approach with main focus on behavioral activation and cognitive restructuring and are carried out by licensed cognitive-behavioral psychotherapists receiving weekly to bi-weekly supervision.

In both conditions, depressive symptoms are monitored with the Patient Health Questionnaire depression module (PHQ-9) at the personal session at baseline and the fourth and eighth telephone sessions. Additionally, psychotherapists complete non-standardized assessments regarding general progress and therapeutic alliance after each session. Decisions about further treatment are to be supported by monitoring results: If symptoms are reduced by at least 20% from baseline to the fourth telephone session, the following sessions are to be stretched to a bi-weekly frequency; if not, continued weekly sessions are recommended. If the PHQ-9-score lies under the cut-off point of 5 by the eighth session, patients are to continue with maintenance therapy. If the PHQ-9-score remains above the cut-off point, transfer into a higher-intensity treatment is recommended. For those patients receiving maintenance therapy, a further monitoring at the end of maintenance therapy is performed and patients above the PHQ-9 cut-off score are also recommended to transfer to a higher-intensity treatment. In case of acute suicidality, emergency measures are carried out: e.g. additional psychiatric treatment in an in- or outpatient setting. Psychotherapists contact the patients' general physicians at begin and end of treatment, as well as on other occasions if necessary. Psychotherapists facilitate transferrals to other mental health care specialists within the stepped care project if necessary.

Patients in the study condition "Tel-PT including mail" receive a one-page letter from their psychotherapist after every telephone session. The letter contains motivational messages as well as a summary of the homework planned during the session and a reminder of the appointment made for the next session. The letters will usually be received by patients approximately two to three days after the telephone session and are meant to refresh memory of and motivation for the planned assignments.

Patients in the study condition "Tel-PT without mail" receive no letters from their psychotherapist.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild or moderate depression
* sufficient knowledge of German language
* health situation that allows questionnaire completion

Exclusion Criteria:

* insufficient knowledge of German language
* health condition not allowing questionnaire completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in depression symptom severity (PHQ-D-9) | Baseline, approximately 3 months (end of treatment)
  Change in patient-rated depression symptom severity: Patient Health Questionnaire 9, German version (PHQ-D-9; Löwe, Zipfel & Herzog, 2002)

SECONDARY OUTCOMES:
Patient-rated acceptance of intervention | Approximately 3 months (end of treatment)
  Patients rate their acceptance of the intervention using non-standardized items.
Need for further, more intensive treatment for depression (therapist-rated) | Approximately 3 months (end of treatment)
  The treating psychotherapist rates the necessity of stepping the patient up to a further, more intensive treatment for depression.
Premature dropout from treatment | Approximately 3 months (end of treatment)
  The rate at which patients drop out from treatment prematurely.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Watzke, Prof. Dr., Study Director — Centre for Psychosocial Medicine, Department of Medical Psychology, University Medical Centre Hamburg-Eppendorf , Hamburg, Germany
Locations (1):
- Centre for Psychosocial Medicine, Department of Medical Psychology, University Medical Centre Hamburg-Eppendorf, Hamburg, Hamburg, Germany